CLINICAL TRIAL: NCT06127407
Title: A Phase 3, Multicenter, Double-blind, Randomized, Placebo-controlled Study of Ivosidenib in Participants ≥18 Years of Age With Locally Advanced or Metastatic Conventional Chondrosarcoma With an IDH1 Mutation, Untreated or Previously Treated With 1 Systemic Treatment Regimen
Brief Title: Ivosidenib in Participants With Locally Advanced or Metastatic Conventional Chondrosarcoma Untreated or Previously Treated With 1 Systemic Treatment Regimen
Acronym: CHONQUER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Servier Bio-Innovation LLC (Industry)
Collaborators: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CL3-95031-007
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Locally Advanced or Metastatic Conventional Chondrosarcoma With an IDH1 Mutation, Untreated or Previously Treated With 1 Systemic Treatment Regimen
Keywords: Conventional chondrosarcoma; IDH1; ivosidenib; locally advanced; metastatic
MeSH Terms: conditions — Neoplasm Metastasis | interventions — ivosidenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ivosidenib (Experimental): Taken continuously until BICR-confirmed disease progression, unacceptable toxicity, confirmed pregnancy, death, withdrawal of consent, lost to follow-up, or the Sponsor ends the study (estimated average treatment duration of two years).
  Interventions: Drug: Ivosidenib 500mg
- Placebo (Placebo Comparator): Taken continuously until BICR-confirmed disease progression, unacceptable toxicity, confirmed pregnancy, death, withdrawal of consent, lost to follow-up, or the Sponsor ends the study (estimated average treatment duration of two years). Participants randomized to the placebo arm who experience BICR-confirmed disease progression and meet the crossover eligibility criteria will be given the opportunity to cross over and receive ivosidenib.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivosidenib 500mg — Provided as tablets, taken orally as two 250mg tablets once daily.
  Arms: Ivosidenib
Drug: Placebo — Provided as tablets, taken orally once daily.
  Arms: Placebo

SUMMARY:
Study CL3-95031-007 (CHONQUER) is a Phase 3, international, multicenter, double-blind, randomized, placebo-controlled study of orally administered ivosidenib. Participants are required to have a histopathological diagnosis consistent with isocitrate dehydrogenase-1 (IDH1) gene-mutated, locally advanced or metastatic conventional chondrosarcoma Grades 1, 2, or 3 and not eligible for curative resection. IDH1 mutant status will be determined during pre-screening/screening phase. Participant must have radiographic progression/recurrence of disease according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1) and have received 0 to 1 prior systemic treatment regimen in the advanced/metastatic setting for conventional chondrosarcoma. The primary endpoint is progression-free survival (PFS) in Grades 1 and 2 participants. Key secondary endpoints are PFS in all randomized participants, overall survival (OS) in Grades 1 and 2 participants, and OS in all randomized participants.

Participants who meet enrollment criteria will be randomized 1:1 to receive oral ivosidenib 500mg once daily, or a matching placebo once daily.

ELIGIBILITY:
Inclusion Criteria:

* Have a histopathological diagnosis (fresh or banked tumor biopsy sample collected within the last 3 years) consistent with locally advanced or metastatic conventional chondrosarcoma Grades 1, 2, or 3 and not eligible for curative resection.
* Have at least one BICR-confirmed measurable lesion as defined by RECIST v1.1. Participants who have received prior radiation therapy are eligible provided measurable disease falls outside of the treatment field or within the field and has shown ≥20% growth in size since post-treatment assessment.
* Have received 0 or 1 prior systemic treatment regimen in the advanced/metastatic setting for chondrosarcoma.
* Have radiographic progression/recurrence of disease according to RECIST v1.1 defined as:

  1. Radiographic progression of disease (local and/or distant) documented by 2 imaging assessments performed no more than 6 months (±2 weeks) apart within 12 months before randomization.

     OR
  2. Any recurrence of disease (local and/or distant) after complete surgical resection and documented by imaging within 6 months (±2 weeks) before randomization.
* Have documented IDH1 gene-mutated disease (from a fresh tumor biopsy or the most recent banked tumor tissue available that was sourced from either a primary or metastatic tumor lesion) based on central laboratory testing (R132C/L/G/H/S mutation variants tested)
* Have recovered from any clinically relevant sequelae and toxic effects of any prior surgery, radiotherapy, or other therapy intended for the treatment of cancer.

Exclusion Criteria:

* Are unable to swallow oral medication.
* Pregnant or lactating women.
* Are participating in another interventional study at the same time; participation in noninterventional registries or epidemiological studies is allowed.
* Have received prior therapy with an IDH1 inhibitor
* Have received systemic anticancer therapy <2 weeks prior to randomization (for investigational or immune-based anticancer therapy <4 weeks).
* Have received radiotherapy <2 weeks prior to randomization.
* Have known symptomatic brain metastases requiring steroids >10 mg per day prednisone (or equivalent). Participants with previously diagnosed brain metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to randomization, have discontinued or reduced corticosteroid treatment <=10 mg per day for these metastases for at least 4 weeks and have radiographically stable disease of brain lesions for at least 3 months prior to randomization.
* Have a history of another primary cancer, with the exception of: a) curatively resected non-melanoma skin cancer; b) curatively treated carcinoma in situ; or c) pT1-2 prostatic cancer Gleason score <6 or d) participant is free of other primary solid or liquid tumor for ≥ 1 year prior to the start of study treatment and, in the opinion of the Investigator, the disease will not affect participant's outcome in the setting of current chondrosarcoma diagnosis.
* Have had major surgery within 4 weeks prior to randomization.
* Have significant active cardiac disease within 6 months prior to randomization, including New York Heart Association (NYHA) Class III or IV congestive heart failure; myocardial infarction; unstable angina; and/or stroke.
* Have LVEF <40% by ECHO scan (or by other methods according to institutional practice) obtained within 28 days prior to randomization.
* Have a heart-rate corrected QT interval (using Fridericia's formula) (QTcF) ≥ 450 msec or other factors that increase the risk of QT prolongation or arrhythmic events (eg, heart failure, hypokalemia, family history of long QT interval syndrome). Participants with a bundle branch block combined with a prolonged QTcF interval may be permitted based on local cardiology assessment.
* Have known medical history of progressive multifocal leukoencephalopathy (PML).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2030-11-26 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) based on Blinded Independent Central Reviewer (BICR) assessment in Grade 1 and Grade 2 participants | Up to approximately 31 months
  From randomization until BICR confirmed progressive disease or death due to any cause, whichever occurs first

SECONDARY OUTCOMES:
PFS based on BICR assessment in all randomized participants | Up to approximately 31 months
  From randomization until BICR confirmed progressive disease or death due to any cause, whichever occurs first
Overall survival (OS) in Grade 1 and Grade 2 participants | Up to 5 years
  From randomization until death
OS in all randomized participants | Up to 5 years
  From randomization until death
PFS based on Investigator assessment in Grade 1 and Grade 2 participants | Up to approximately 31 months
  From randomization until BICR confirmed progressive disease or death due to any cause, whichever occurs first
PFS based on Investigator assessment in all randomized participants | Up to approximately 31 months
  From randomization until BICR confirmed progressive disease or death due to any cause, whichever occurs first
Objective response (OR) (confirmed complete response(CR) or confirmed partial response (PR)) of anti-tumor activity (using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1) in Grade 1 and Grade 2 participants | Up to approximately 31 months
  From randomization until confirmed CR or PR
OR (confirmed CR or confirmed PR) of anti-tumor activity (using RECIST v1.1) in all randomized participants | Up to approximately 31 months
  From randomization until confirmed CR or PR
Duration of response (DOR) in Grade 1 and Grade 2 participants | Up to approximately 31 months
  The time from date of first documented confirmed CR or confirmed PR to date of first documented disease progression or death due to any cause.
DOR in all randomized participants | Up to approximately 31 months
  The time from date of first documented confirmed CR or confirmed PR to date of first documented disease progression or death due to any cause.
Time to response (TTR) in Grade 1 and Grade 2 participants | Up to approximately 31 months
  The time from the date of randomization to date of first documented confirmed complete response (CR) or confirmed partial response (PR).
TTR in all randomized participants | Up to approximately 31 months
  The time from the date of randomization to date of first documented confirmed complete response (CR) or confirmed partial response (PR).
Disease control (DC) confirmed CR, confirmed PR, or stable disease (SD)) in Grade 1 and Grade 2 participants | Through the end of the study (a maximum of 5 years after the study start)
DC (confirmed CR, confirmed PR, or SD) in all randomized participants | Through the end of the study (a maximum of 5 years after the study start)
Duration of disease control (DoDC) in Grade 1 and Grade 2 participants | Through the end of the study (a maximum of 5 years after the study start)
DoDC in all randomized participants | Through the end of the study (a maximum of 5 years after the study start)
Number of Adverse Events (AEs) | Through the Safety Follow-up Visit (28-33 days after discontinuation of treatment)
Number of Serious Adverse Events (SAEs) | Through the Safety Follow-up Visit (28-33 days after discontinuation of treatment)
Number of Adverse Events of Special Interest (AESIs) | Through the Safety Follow-up Visit (28-33 days after discontinuation of treatment)
Number of Adverse Events (AEs) leading to discontinuation, treatment interruption, and dose reduction | Through the Safety Follow-up Visit (28-33 days after discontinuation of treatment)
European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) score | Through the Safety Follow-up Visit (28-33 days after discontinuation of treatment)
  The EORTC-QLQ-C30 contains 30 items across 5 functional scales, 9 symptom scales and a global health status. Raw scores are converted to scales ranging from 0 - 100. For the functional scales and global health status, the higher score represents the better functioning or global health status; for the symptom scales, the higher score represents an increase in symptoms.
European Quality of Life 5 Dimensions 5 Level (EQ-5D-5L) score | Through the Safety Follow-up Visit (28-33 days after discontinuation of treatment)
  The 5-level EQ-5D-5L scores range from 5 to 25 with a higher number representing a worse health status.
Patient-Reported Outcomes Measurement Information System (PROMIS) score | Through the Safety Follow-up Visit (28-33 days after discontinuation of treatment)
  The PROMIS Item Bank v1.0 Physical Function with Mobility Aid - Short Form questionnaire score ranges from 1 "Unable to do" to 5 "Can do without a problem" for each capability.
Ivosidenib concentration in plasma | Through the end of the study (a maximum of 5 years after the study start)
2-hydroxyglutarate (2-HG) concentration in plasma | Through the end of the study (a maximum of 5 years after the study start)

CONTACTS AND LOCATIONS:
Locations (113):
- United States (22):
  - Usc Norris Comprehensive Cancer Center, Los Angeles, California
  - Sarcoma Oncology Research Center, Santa Monica, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Mayo Clinic - Jacksonville, Fl, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - University of Iowa Hospitals & Clinics- Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic - Rochester, Mn, Rochester, Minnesota
  - The Washington University, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health & Science University Knight Cancer Institute, Portland, Oregon
  - University of Pittsburgh Medical Center-Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The Univeristy of Texas Md Anderson Cancer Center, Houston, Texas
- Australia (5):
  - Flinders Medical Centre, Bedford Park
  - Chris O'Brien Lifehouse, Camperdown
  - St Vincent'S Hospital Melbourne, Fitzroy
  - Sir Charles Gairdner Hospital, Nedlands
  - Princess Alexandra Hospital, Woolloongabba
- Belgium (3):
  - Cliniques Universitaires St. Luc, Brussels
  - U.Z. Gent, Ghent
  - Centre Multidisciplinaire de Oncologie Medicale, Liège
- Brazil (11):
  - Liga Norte Riograndense Contra O Cancer, Natal, Rio Grande do Norte
  - Hospital de Amor - Barretos, Barretos
  - Hospital Das Clínicas Da Ufmg, Belo Horizonte
  - CIONC, Curitiba
  - Cepon - Centro de Pesquisas Oncologicas, Florianópolis
  - Fundação Amaral Carvalho - Jaú/ Sp, Jaú
  - Instituto Nacional Do Câncer - Inca, Rio de Janeiro
  - Icesp - Instituto Do Câncer Do Estado de São Paulo, São Paulo
  - Impar Serviços Hospitalares S.A. - Hospital Nove de Julho, São Paulo
  - Hospital A C Camargo, São Paulo
  - Hospital Albert Einstein, São Paulo
- Canada (3):
  - Alberta Health Services, Calgary, Alberta
  - University Health Network, Toronto, Ontario
  - Muhc Glen Site, Montreal, Quebec
- China (10):
  - The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Shanghai Changzheng Hospital, Shang'ai, Shanghai Municipality
  - Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - West China Hopital of Sichuan University, Chengdu, Sichuan
  - The Second Affiliated Hospital Zhejiang University School of Medical, Hangzhou, Zhejiang
  - Beijing Cancer Hospital, Beijing
  - Beijing Jishuitan Hospital, Beijing
  - Henan Cancer Hospital, Guangzhou
- Denmark (2):
  - Aarhus Universitetshospital, Aarhus
  - Herlev & Gentofte Hospital, Herlev
- France (8):
  - Institut Bergonié, Bordeaux
  - Centre Oscar Lambret, Lille
  - Hôpital Léon Bérard, Lyon
  - Hopital de La Timone, Marseille
  - Hôpital Cochin, Paris
  - INSTITUT de CANCEROLOGIE de l'Ouest, Saint-Herblain
  - Iuct-Oncopole Institut Universitaire Du Cancer, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (8):
  - Helios Klinikum Bad Saarow, Bad Saarow
  - Charite Universitatsmedizin, Berlin
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsmedizin Mannheim (Umm), Mannheim
  - Lmu Klinikum, München
  - Ukm - Sarkom-Zentrum, Münster
  - Universitaetsklinikum Ulm, Ulm
- Italy (8):
  - Irccs Istituto Ortopedico Rizzoli, Bologna
  - Irccs Fondazione Istituto Nazionale Dei Tumori, Milan
  - San Luigi Gonzaga University Hospital of Turin, Orbassano
  - Istituto Oncologico Veneto Iov - Irccs, Padua
  - Aou Policlinico Paolo Giaccone, Palermo
  - Ospedale Santo Stefano, Prato
  - Policlinico Universitario Campus Biomedico, Roma
  - Istituti Fisioterapici Ospitalieri (Ifo) - Istituto Nazionale Tumori Regina Elena (Ire), Roma
- Japan (11):
  - Hokkaido Cancer Center, Sapporo, Hokkaido
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Nagoya University Hospital, Shōwaku, Nagoya-shi, Aichi
  - Niigata University Medical and Dental General Hospital, Chūōku, Niigata City
  - Oita University Hospital, Yufu-Shi, Oita Prefecture
  - Osaka International Cancer Institute, Chūōku, Osaka-shi, Osaka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Fukushima Medical University Hospital, Fukushima
  - Kyushu University Hospital, Higashi
  - Cancer Institute Hospital of Jfcr, Koto-Ku, Tokyo
  - Okayama University Hospital, Okayama
- Netherlands (3):
  - Universitair Medisch Centrum Groningen (Umcg), Groningen
  - Leids Universitair Medisch Centrum, Leiden
  - Radboud Umc, Nijmegen
- Pan American Center For Oncology Trials, LLC, Rio Piedras, Puerto Rico
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (7):
  - Hospital Universitario Valle de Hebrón - Vhio, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital de Bellvitge - Ico, L'Hospitalet de Llobregat
  - Hospital General Universitario Gregorio, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Y Politecnico La Fe, Valencia
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (5):
  - Western General Hospital, Edinburgh
  - Royal Marsden Hospital, London
  - UCLH, London
  - Christie Hospital, Manchester
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorization in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com/

REFERENCES:
- [Derived] Tap WD, Cote GM, Burris H, Gore L, Elias A, Beeram M, Conley AP, Gianolio DA, Qu Z, Pandya S, Trent JC. Phase I Study of the Mutant IDH1 Inhibitor Ivosidenib: Long-term Safety and Clinical Activity in Patients with Conventional Chondrosarcoma. Clin Cancer Res. 2025 Jun 3;31(11):2108-2114. doi: 10.1158/1078-0432.CCR-24-4128. PMID 40100120
- See also: CHONQUER Study Website — https://chonquer.com/en-us/